CLINICAL TRIAL: NCT02630420
Title: Combination of Cetuximab & MWT Inhibitor Savolitinib in the Treatment of Ras Wild-Type Colorectal Cancer
Brief Title: Cetuximab and Savolitinib Treatment of Ras Wild-Type Colorectal Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study never officially funded and therefore never began.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1502015402
Record Dates: First submitted 2015-12-01; First posted 2015-12-15 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cetuximab and savolitinib (Experimental): Following assessment in Part 1 of dose-limiting toxicity and maximum tolerated dose, this drug combination will be administered in Part 2 of the study to assess safety, tolerability, response rate, and progression-free survival.
  Interventions: Drug: cetuximab and savolitinib

INTERVENTIONS:
Drug: cetuximab and savolitinib — Dosage of combined cetuximab and savolitinib will be determine in Part 1 of the study, Part 2 will use the findings of Part 1 to further assess safety and to assess efficacy of this drug combination.

SUMMARY:
Two-part phase 1B clinical trial combining cextuximab and savolitinib for treating Ras wild-type colorectal cancer (CRC). Part 1 will assess the safety and tolerability of this drug combination and will include patients with squamous cell carcinoma of the head and neck cancer, as well as patients with CRC. Part 2 of the study, the focus of this registration, will obtain further safety data for the combination of cextuximab and savolitinib and will look at the efficacy of cextuximab and savolitinib in Ras wild-type mCRC that was previously treated and relapsed on cetuximab or panitumumab.Correlative studies will examine tumor and blood specimens for mechanisms of anti-EGFR resistance and response to MET inhibition.

ELIGIBILITY:
Inclusion Criteria, Part 1:

1. Progressive metastatic or unresectable CRC or SCCHN.
2. Prior therapy with cetuximab or panitumumab. Cetuximab and panitumumab could have been used either alone or in combination with other agents.
3. If patients were treated with cetuximab in the past, they must have been able to tolerate full doses of cetuximab without dose modifications for toxicity.
4. ECOG performance status 0-2.
5. Life expectancy of at least 3 months.
6. Patient with adequate organ function:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Hemoglobin ≥ 9 g/dL
   * Platelets (PLT) ≥ 100 x 109/L
   * AST/ALT ≤ 2.5 x ULN (≤ 5 x ULN in case of liver metastases)
   * GGT < 3 x ULN (< 5 x ULN in case of liver involvement)
   * Bilirubin ≤ 1.5 x ULN
   * Albumin ≥ 3 g/dL
   * Serum creatinine ≤ 1.5 x institutional ULN (Cockcroft and Gault formula)
7. Adequate contraception if applicable.
8. Ability to take oral medication in the opinion of the investigator.
9. Patient able and willing to comply with study procedures as per protocol, including the biopsy at the time of study enrollment.
10. Patient able to understand and willing to sign and date the written voluntary informed consent form (ICF) at screening visit prior to any protocol-specific procedures.

Inclusion Criteria, Part 2:

1. Histologically confirmed stage IV colon cancer (AJCC 7th edition) that has progressed after at least one line of standard therapy.
2. Presence of measurable disease per RECIST criteria on imaging studies at the time of trial enrollment.
3. Prior therapy with cetuximab or panitumumab containing regimen and disease progression within 3 months of last dose of cetuximab or panitumumab. Anti-EGFR antibodies could have been used either alone or in combination with other agents.
4. Subjects should be off other disease directed treatments for at least 4 weeks prior to treatment initiation on this study.
5. Absence of K-Ras or N-Ras mutations using extended Ras profiling.
6. ECOG performance status 0-2.
7. Life expectancy of at least 3 months.
8. Patient able to receive adequate oral nutrition of ≥ 1500 calories per day and free of significant nausea and vomiting
9. Patient with adequate organ function:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Hemoglobin ≥ 9 g/dL
   * Platelets (PTL) ≥ 100 x 109/L
   * AST/ALT ≤ 2.5 x ULN (≤ 5 x ULN in case of liver metastases)
   * Bilirubin ≤ 1.5 x ULN
   * Albumin ≥ 3 g/dL
   * Serum creatinine ≤ 1.5 x institutional ULN (Cockcroft and Gault formula)
10. Adequate contraception if applicable.
11. Ability to take oral medication in the opinion of the investigator.
12. Patient able and willing to comply with study procedures as per protocol, including a tumor biopsy within 28 days of treatment initiation.
13. Patient able to understand and willing to sign and date the written voluntary informed consent form at screening visit prior to any protocol-specific procedures.

Exclusion Criteria (Parts 1 and 2):

1. Previous treatment with MET inhibitor or anti-MET antibody (e.g. foretinib, crizotinib, cabozantinib, onartuzumab).
2. Patients with previous hypersensitivity to cetuximab (Grade 2 or higher, unless controlled to < Grade 2 with prophylactic measures on subsequent exposures).
3. Active dermatological condition requiring treatment with associated grade 2 or higher skin toxicity. Dermatological condition controlled with treatment with maximum of grade 1 skin toxicity will be allowed for study enrollment.
4. Symptomatic brain metastases requiring treatment.
5. Other active malignancy within the last 3 years (except for non-melanoma skin cancer or a non-invasive/in situ cancer).
6. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
7. Persistent toxicities CTCAE grade 2 or higher, with the exception of alopecia, caused by previous cancer therapy.
8. Pregnancy or breast feeding.
9. Current therapy with other investigational agents or participation in another clinical study.
10. History of allergic reactions attributed to compounds of similar chemical or biologic composition to savolitinib.
11. Major surgery within 28 days or minor surgery within 14 days of the start of the study treatment, except for tumor biopsy.
12. Radiotherapy less than two weeks prior to the start of the study treatment
13. Significant current or recent (< 14 days) gastrointestinal disorders with diarrhea as a major symptom, e.g. Crohn's disease, malabsorption, or CTCAE grade > 2 diarrhea of any etiology.
14. Psychological, familial, or sociological condition potentially hampering compliance with the study protocol and follow-up schedule.
15. Involvement in the planning and/or conduct of the study.
16. Previous enrolment in the present study.
17. Acute or chronic liver or pancreatic disease.
18. Use of strong inducers or inhibitors of CYP3A4 or strong inhibitors of CYP1A2 within 2 weeks before the first dose of study treatment (3 weeks for St John's Wort).

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability based on regular clinical assessment and NCI Common Terminology Criteria for Adverse Events | start of treatment to 3 years from treatment initiation

SECONDARY OUTCOMES:
Response to treatment measured by RECIST (Response Evaluation Criteria in Solid tumors) criteria | start of treatment to disease progression/recurrence, up to 3 years
Progression free survival | start of treatment to disease progression, up to 3 years

OTHER OUTCOMES:
HGF/MET pathway activation as a predictor of response to therapy. | 3 years from start of treatment
  HGF/MET pathway activation will be assessed by MET mutation or amplification in tumor or plasma, or MET/HGF protein expression in tumor tissue.
Genetic aberrations, assessed by next generation sequencing, as predictors of sensitivity/resistance to treatment. | 3 years from start of treatment
Changes in HGF/MET pathway activation over the course of the disease measured by comparing archival, baseline and progression samples. | 3 years from start of trial
Changes in genetic aberrations over the course of the disease by comparing archival, baseline and progression samples. | 3 years from start of trial

CONTACTS AND LOCATIONS:
Overall Officials: Stacey M Stein, MD, Principal Investigator — Yale University